CLINICAL TRIAL: NCT06198530
Title: Effectiveness of Nurse-led Clinics Training Program on Mild Cognitive Impairment Patients: a Randomized Controlled Trial Protocol
Brief Title: Nurse-led Clinics Training Program on Mild Cognitive Impairment Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021029
Record Dates: First submitted 2023-08-09; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-08

CONDITIONS: Mild Cognitive Impairment
Keywords: nurse-led clinics; computerized cognitive training; randomized controlled clinical trial
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training; Home Care Services

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Radiologists, statisticians, and neuropsychologists who measure the outcomes will be blinded to the randomization status. Blinding will also be maintained for data management, outcome assessment, and data analysis. Participants and therapists cannot be blinded to the intervention they receive or provide.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cognitive training in NLCs (Active Comparator): computerized cognitive training (CCT) was given twice a week during 1-6 months and once a week during 7-12 month in nursing clinic. There is 60 minutes at a time. All the patients were capable of performing the training under the guidance of advanced practicing nurses (APNs). At the same time, according to the caregivers' feedback, APNs will give them the desired care guidance.
  Interventions: Behavioral: cognitive training in NLCs
- cognitive training in home (Active Comparator): CCT was given four times a week during 1-6 months and twice a week during 7-12 month in nursing clinic. There is 30 minutes at a time. Nurses teach patients to acquire and carry out CCT at home during hospitalization. Nurses set the daily reminder function at 9:00am through training system. The data results of each training will be automatically stored in the personal information database in the cloud. And, a training report will be generated, including training difficulty, training results and training time. Nurses can examine patients' training through the cloud.
  Interventions: Behavioral: cognitive training in home
- cognitive training in tradition (Placebo Comparator): the Home Cognitive Training Manual for Alzheimer's Disease compiled by our research team was distributed. And, the patients and their families were given detailed health education on the definition, clinical manifestations, drug and non-drug treatment, home nursing, the significance of cognitive training and the methods of cognitive training. Meanwhile, we established connection with patients for later follow-up
  Interventions: Behavioral: cognitive training in tradition

INTERVENTIONS:
Behavioral: cognitive training in NLCs — In the nurse-led clinics(NLCs) training group, CCT was given twice a week during 1-6 months and once a week during 7-12 month in nursing clinic. There is 60 minutes at a time.
  Arms: cognitive training in NLCs
Behavioral: cognitive training in home — In the home-based training group, CCT was given four times a week during 1-6 months and twice a week during 7-12 month in nursing clinic. There is 30 minutes at a time. Nurses teach patients to acquire and carry out CCT at home during hospitalization. Nurses set the daily reminder function at 9:00am through training system.
  Arms: cognitive training in home
Behavioral: cognitive training in tradition — In the traditional training group, the Home Cognitive Training Manual for Alzheimer's Disease compiled by our research team was distributed.
  Arms: cognitive training in tradition

SUMMARY:
This trail is the first study to test the efficacy of nurse-led clinics cognitive training on mild cognitive impairment (MCI) patients using a single-blind, randomized controlled trial design. The investigators hypothesize that nurse-led clinics cognitive training can (a)decelerate or ameliorate cognitive decline, (b)ameliorate anxiety and depressive symptoms, (c)increase the quality of life for both patients and family members, (d)improve the ability of daily life, (e)reduce the incidence of agitation.

DETAILED DESCRIPTION:
Introduction: Globally, nurse-led clinics(NLCs) have been developed to serve and follow up on patients who have just been discharged from the hospital. NLCs cognitive training program as a potentially effective and promising treatment for MCI patients.

Methods: The study is a single-blind, randomized-controlled trial. Eligible patients need to be diagnosed as MCI. Participants will be randomized into either a NLCs training group or a home-based training group. Both groups will undergo total 72hour across 12 months. The outcome measures will be assessed at baseline, at the 6 months and 12 months during the intervention. The primary outcome is global cognitive function, assessed by the 30-item the Mini-Mental State Examination (MMSE), and the secondary outcomes include changes in other neuropsychological assessments and in result of resting electroencephalography (EEG) .

Results: The trial is currently ongoing, and it is anticipated that recruitment will be completed in June 2025.

Discussion: This trial will evaluate the efficacy and safety of NLCs cognitive training in patients with MCI, and further explore the potential mechanisms by analyzing teh results of neuropsychological assessments and EEG.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with informed consent;
* Literate Han Chinese, above the age of 18;
* At least 6 years of education;
* Neither normal nor demented according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, with a Clinical Dementia Rating(CDR) ≥0.5 on at least one domain and a global score ≤0.5; a Mini-Menta State Examination score ≥20 (primary school), or ≥24 (junior school or above).
* having normal vision and hearing with/without corrective devices.

Exclusion Criteria:

* Severe aphasia, physical disabilities, or any other factor that might preclude completion of neuropsychological testing.
* Clinically significant gastrointestinal, renal, hepatic, respiratory, infectious, endocrine, or cardiovascular system disease; cancer; alcoholism; drug addiction.
* Illnesses affecting mobility or are unable to accept assessments or interventions that are required in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 96 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Mini-Mental State Examination (MMSE) | From baseline to the 6-month and 12-month after intervention
  The intervention will be assessed by the MMSE in which scores range from 0 to 30, with higher scores representing better general cognitive performance.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) | From baseline to the 6-month and 12-month after intervention
  Montreal Cognitive Assessment in which scores range from 0 to 30, with higher scores representing better general cognitive performance.
Change in World Health Organization-University of California-Los Angeles Auditory Verbal Learning Test (WHO-UCLA AVLT) | From baseline to the 6-month and 12-month after intervention
  World Health Organization-University of California-Los Angeles Auditory Verbal Learning Test , which scores range from 0 to 45 will be used to assess memory function in which scores range from 0 to 45, with a higher value representing a better outcome.
Change in Boston Naming Test (BNT) | From baseline to the 6-month and 12-month after intervention
  Boston Naming Test in which scores range from 0 to 30 will be used to assess language performance, specifically visual naming ability.
Change in Instrumental activities of daily living(IADL) | From baseline to the 6-month and 12-month after intervention
  Instrumental activities of daily living in which scores range from 0 to 24 were defined as being whether able to complete Instrumental activity ability.
Change in the barthel index（BI） | From baseline to the 6-month and 12-month after intervention
  the barthel index in which scores range from 0 to 100 were defined as being whether able to complete basic activity ability.
Change in Hamilton Anxiety rating scale(HARS) | From baseline to the 6-month and 12-month after intervention
  Hamilton Anxiety rating scale in which scores range from 0 to 56 measures14 items, adopt Likert5 level score, the higher the score according to the more serious the degree of anxiety
Change in Geriatric depression scale(GDS) | From baseline to the 6-month and 12-month after intervention
  Geriatric depression scale measures 30 items，in which scores range from 0 to 30. The higher the score according to the more serious the degree of depression
Change in Cohen-Mansfield Agitation Inventory (CMAI) | From baseline to the 6-month and 12-month after intervention
  The Cohen-Mansfield Agitation Inventory measures 29 agitated or aggressive behaviors. The frequency of each symptom is rated on a seven-point scale (1-7) ranging from "never" to "several times an hour."the scores range from 29 to 203. The higher the score according to the more serious the degree of agitation
Change in Neuropsychiatric Inventory(NPI) | From baseline to the 6-month and 12-month after intervention
  The Neuropsychiatric Inventory consists of 12 items that are assayed with questions, subquestions, and ratings of frequency and severity. the scores range from 0 to 144. The higher the score according to the more serious the degree of mental and behavioral abnormalities
Change in Zarit caregiver burden interview (ZBI) | From baseline to the 6-month and 12-month after intervention
  Zarit caregiver burden interview contains 29 items on a four-point Likert scale, will be used to assess the burden of caregivers.
Change in Resting EEG | From baseline to the 6-month and 12-month after intervention
  EEG was acquired using a 32-conductor electrode cap and amplifier (BioSemi, Amsterdam, Netherlands) with a 2048-Hz sampling rate. To reduce interference during signal acquisition, we ensured that the electrode resistance was<5 kΩ. During data collection, the participants were seated in a comfortable chair, relaxed, refrained from speech or voluntary movements, and kept their eyes closed. The eyes-closed state was recorded for 5 min, and the data were stored on a computer for offline analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Background] Sanford AM. Mild Cognitive Impairment. Clin Geriatr Med. 2017 Aug;33(3):325-337. doi: 10.1016/j.cger.2017.02.005. Epub 2017 May 17. PMID 28689566
- [Background] Jia L, Du Y, Chu L, Zhang Z, Li F, Lyu D, Li Y, Li Y, Zhu M, Jiao H, Song Y, Shi Y, Zhang H, Gong M, Wei C, Tang Y, Fang B, Guo D, Wang F, Zhou A, Chu C, Zuo X, Yu Y, Yuan Q, Wang W, Li F, Shi S, Yang H, Zhou C, Liao Z, Lv Y, Li Y, Kan M, Zhao H, Wang S, Yang S, Li H, Liu Z, Wang Q, Qin W, Jia J; COAST Group. Prevalence, risk factors, and management of dementia and mild cognitive impairment in adults aged 60 years or older in China: a cross-sectional study. Lancet Public Health. 2020 Dec;5(12):e661-e671. doi: 10.1016/S2468-2667(20)30185-7. PMID 33271079
- [Background] Wang Q, Zhang Z, Li L, Wen H, Xu Q. Assessment of cognitive impairment in patients with Parkinson's disease: prevalence and risk factors. Clin Interv Aging. 2014 Feb 12;9:275-81. doi: 10.2147/CIA.S47367. eCollection 2014. PMID 24550669
- [Background] Benedict RHB, Amato MP, DeLuca J, Geurts JJG. Cognitive impairment in multiple sclerosis: clinical management, MRI, and therapeutic avenues. Lancet Neurol. 2020 Oct;19(10):860-871. doi: 10.1016/S1474-4422(20)30277-5. Epub 2020 Sep 16. PMID 32949546
- [Background] How Many People Have Dementia and What Is the Cost of Dementia Care? Alzheimer's Society.2019. URL: https://www. alzheimers.org.uk/about-us/policy-and-influencing/dementia-scale-impact-numbers.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT06198530/Prot_SAP_000.pdf